CLINICAL TRIAL: NCT00812136
Title: Using Parent Mentors to Improve Asthma Care for Urban Minority Children
Brief Title: Parent Mentor Asthma Study
Acronym: PMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: PMA-102008-001; NCT00800020 (obsolete NCT alias)
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Asthma
Keywords: Using Parent Mentors to Improve Asthma Care for Urban Minority Children
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Using Parent Mentors to Improve Asthma Care for Urban Minority Children

SUMMARY:
Asthma disproportionately affects minorities, but few studies have evaluated interventions to improve asthma outcomes in minority children.The purpose of the study is to determine whether Parent Mentors (PMs) are more effective than traditional asthma care in reducing minority children's asthma morbidity, costs, and use of services, while increasing families' quality of life and parental self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* The child was 2-18 years old
* African-American or Latino race/ethnicity for the child (by parental identification)
* Primary residence in a Milwaukee zip code
* ED or inpatient ward admission with a primary diagnosis of asthma.

Exclusion Criteria:

* Significant co-morbidity, including other pulmonary conditions, cardiac pathology, renal abnormalities, diabetes mellitus, epilepsy, and other co-morbidities that might lead to ED visits or hospitalizations, and current enrollment in a case management, intervention, or outreach program for childhood asthma management.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gruchalla, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center

REFERENCES:
- [Derived] Flores G, Bridon C, Torres S, Perez R, Walter T, Brotanek J, Lin H, Tomany-Korman S. Improving asthma outcomes in minority children: a randomized, controlled trial of parent mentors. Pediatrics. 2009 Dec;124(6):1522-32. doi: 10.1542/peds.2009-0230. PMID 19948624